CLINICAL TRIAL: NCT01028274
Title: Clinical Trial to Assess the Safety and Efficacy of a Combination Red Yeast Rice and Omega-3 (EPA+DHA) to Reduce LDL Cholesterol and Triglyceride Levels in Hypercholesterolemic and Hypertriglyceridemic Subjects.
Brief Title: Safety and Efficacy of a Natural Health Product in Reducing Cholesterol and Triglyceride Levels.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordic Pharma, USA (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NN-91109; NHPD145265
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: LDL Cholesterol; Triglycerides
Keywords: Hypercholesterolemia; Hypertriglyceridemia; Fish Oil; Red Yeast Rice
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia | interventions — Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Investigational Product 1 (Experimental)
  Interventions: Dietary Supplement: Investigational Product 1
- Investigational Product 2 (Experimental)
  Interventions: Dietary Supplement: Investigational Product 2

INTERVENTIONS:
Dietary Supplement: Placebo — Two capsules, twice daily with meals for 12 weeks.
  Other Names: Soybean Oil; Mfr. Product Code: 31237-NNM
  Arms: Placebo
Dietary Supplement: Investigational Product 1 — Two capsules, twice daily with meals for 12 weeks.
  Other Names: Mfr. Product Code: 31214-NNM
  Arms: Investigational Product 1
Dietary Supplement: Investigational Product 2 — Two capsules, twice daily with meals for 12 weeks.
  Other Names: Mfr. Product Code: 31236-NNM
  Arms: Investigational Product 2

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a natural health product among participants with elevated LDL cholesterol and triglyceride levels.

DETAILED DESCRIPTION:
Cardiovascular Disease [CVD] is one of the primary causes of illness, disability and death in Canada and in the United States. Hypercholesterolemia and hypertriglyceridemia are significant risk factors for the development of cardiovascular disease.

The investigational product used in this trial, has been specially formulated to help reduce elevated triglycerides and LDL cholesterol levels, and may provide a natural alternative in the prevention of CVD.

This study is a prospective, 12 week study, where participants will be randomized to receive the treatment, placebo, or a comparator product for a period of 12 weeks. Blood lipids will be analysed at baseline, week 6 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 - 70 years.
* 10-year CAD Risk <10%
* Elevated blood LDL cholesterol in the range of 3.0 to 5.0 mmol/L [equivalent to 117-195 mg/dl].
* have elevated TG levels [1.5/L - 4.0mmol/L, or 134 mg/dl - 356 mg/dl].

Exclusion Criteria:

* Adults aged less than 30, or more than 70 years of age
* Adults with a 10-year CAD risk >10%
* Individuals with a pre-existing disease or illness including: heart disease, diabetes, renal disease or cancer
* Individuals taking CYP3A4 inhibitors [including cyclosporine and danazol].
* Individuals taking Statin medications, including: Atorvastatin [brand names: Lipitor®, Caduet®]

  * Fluvastatin [brand names: Lescol®, Lescol® XL]
  * Lovastatin [brand names: Advicor ®, Altocor ®, Altoprev ®, Mevacor ®]
  * Pravastatin [brand names: Pravachol® , Pravigard® PAC]
  * Rosuvastatin [brand name: Crestor®]
  * Simvastatin [brand names: Vytorin®, Zocor ®]
* Individuals with an allergy to fish and/or fish oil, Vitamin E, red yeast rice, coenzyme Q10, soybean oil or any other ingredient in the investigational product [i.e. capsule constituents]
* Individuals who anticipate, or have planned surgery during the course of the trial
* Individuals who are taking any other natural health products, particularly those containing vitamin K, high levels of vitamin E or Coenzyme Q10 [individuals on a 4-week wash-out of NHPs will be permitted]
* Individuals who have consumed fish oil or another type of omega-3 fatty acid supplement one-month prior-to and/or during the course of the study
* Women who are pregnant or breastfeeding
* Individuals with a history of migraines
* Individuals taking blood thinning, or blood pressure medications
* Individuals who have been diagnosed with statin-induced muscle damage (myopathy)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in LDL levels | 0 weeks, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Reduction in TG levels | 0 weeks, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Laidlaw, Ph.D. Candidate, Study Director — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.; Brad West, ND, Study Chair — Nordic Naturals; Steven Traplin, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Diagnostics Inc., Guelph, Ontario, Canada